CLINICAL TRIAL: NCT02603380
Title: Feasibility Study of a Software Application for Detection and Monitoring of Attentional Deficits in Delirium
Brief Title: Feasibility of a Software App for Testing Inattention in Delirium
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Medical Research Council (Other Government); NHS Lothian (Other Government); University of Glasgow (Other); NHS Greater Glasgow and Clyde (Other); Cambridge Cognition Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: DelApp phase A
Record Dates: First submitted 2015-10-19; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Delirium
Keywords: Delirium; Feasibility study; software application; qualitative
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clinical staff: Clinicians in the Royal Infirmary of Edinburgh.
  Interventions: Other: No intervention
- Patients: Patients in intensive care units and general wards in the Royal Infirmary of Edinburgh.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. No intervention will be given.

SUMMARY:
This qualitative study aims to evaluate the usability of a smartphone application called DelApp. The study will assess usability and acceptability of the software app by asking 40 clinicians to administer the DelApp assessment to consented patient and clinicians. Feedback will be collected through semi-structured interviews with the clinicians. The feedback will be used to optimise the software application in preparation for formal validations studies.

DETAILED DESCRIPTION:
Delirium is an acute, serious syndrome involving abnormalities in attention, arousal and cognition. Delirium affects 1 in 8 hospital patients. Delirium is linked to a higher risk of death, increased length of stay, and substantial patient and carer distress. Despite its massive medical importance, delirium is grossly underdetected, with rates of formal detection of 20% or less.

Investigators previously developed a new neuropsychological test for the objective measurement of inattention in delirium, implemented on a computerised device (Delbox). A prototype software application for smartphones (DelApp) has been developed based on the 'Delbox' tests. Findings from two pilot studies suggest that the DelApp performs well as a method for objectively measuring attention in delirium.

As part of a new programme of work on attentional tests for delirium, formally funded by the Medical Research Council (grant value £1.01M), investigators plan further studies to refine the DelApp before conducting larger scale formal studies. The reasons for doing these additional studies are to: (1) shorten the duration of the DelApp assessment; (2) ask end users (i.e. clinicians) to evaluate the user interface; (3) gather feedback from end users regarding the ease of use of the test; and any other feedback from clinicians and patients; and finally (4) develop the DelApp software application further based on user feedback.

Here investigators propose a preliminary qualitative study to evaluate feasibility of the optimised DelApp test (points 2 and 3). Investigators will assess usability and acceptability by asking 40 clinical staff to administer the DelApp test to consented patients (N=10) and colleagues (approximately N=30). Feedback will be collected from clinicians and patients through semi-structured interviews. The outcomes of this feasibility study will make further optimisation of the app possible, in preparation for formal validation studies.

ELIGIBILITY:
Inclusion Criteria:

* Native or fluent English speaker

  * Capacity to give consent to participate in the study
  * Aged 65 or over

Exclusion Criteria:

* Vision, hearing or speech impairment severe enough to preclude testing and interview.

  * Known or suspected cognitive impairment including dementia
  * Photosensitive epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Royal Infirmary of Edinburgh (RIE) general wards and intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Semi-structured interviews with clinicians and patients to produce a set of recommendations to refine and optimise the DelApp. | Baseline
  Clinicians and patients who have used the DelApp will be interviewed using semi structured interviews.

SECONDARY OUTCOMES:
System usability scale to measure the usability of the DelApp. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: David J Stott, Principal Investigator — University of Glasgow; Elizabeth Wilson, Principal Investigator — NHS Lothian; Timothy Walsh, Principal Investigator — University of Edinburgh; Tara Quasim, Principal Investigator — University of Glasgow; Jonathan Evans, Principal Investigator — University of Glasgow; Christopher Weir, Principal Investigator — University of Edinburgh; Alexander Weir, Principal Investigator — Medical Devices Unit; Stuart Parks, Principal Investigator — Medical Devices Unit; Jenny Barnett, Study Chair — Cambridge Cognition Ltd